CLINICAL TRIAL: NCT03925493
Title: Exercise Prescription in Cardiac Rehabilitation: A Pilot Randomized Controlled Trial
Brief Title: Exercise Prescription in Cardiac Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baystate Medical Center (Other)
Collaborators: Springfield College (Other)
Responsible Party: Principal Investigator, Quinn Pack, MD, MSc, Director, Head of Cardiac Rehabilitation, Principle Investigator, Baystate Medical Center
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BH-19-087
Record Dates: First submitted 2019-04-05; First posted 2019-04-24 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Percutaneous Coronary Intervention; Myocardial Infarction; Coronary Artery Bypass Graft
Keywords: Graded exercise testing; Cardiac rehab; Exercise Prescription; Target heart rate range; RPE
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group Procedures (RPE based exercise) (No Intervention): Patients in the control group will follow standard exercise prescription protocols in CR. Exercise intensity will be guided by the patient's reported rating of perceived exertion (RPE). The modified Borg scale will be used by the patients to determine their RPE. Therefore, a scale of 1-10 will be used. The general goal will be to exercise between intensity level 3 or 4 (i.e. moderate intensity), per current program standards. Based on exercise levels achieved on the first day, patients will be given exercise recommendations for their 2nd session of CR and so forth. As the patients progress in CR, patients will increase their time, intensity, and mode of exercise as appropriate. Exercise progression will be guided by RPE and clinical assessment.
- Exercise Test and Heart Rate Range (Experimental): Patients randomly assigned to this group will complete a graded exercise test (GXT) per standard protocols. The researchers will obtain the patients peak heart rate from this stress test. Obtaining an accurate peak heart rate will allow for the calculation of a target heart rate range (THRR) using the Karvonen formula. Based upon the Karvonen formula, the THRR will be between 60-80% of the patient's heart rate reserve. The Karvonen formula can be calculated as follows ((peak heart rate - resting heart rate) X % intensity (0.6 or 0.8) + resting heart rate)). An example would be: (155 -75) X (.6) + 75) = 123; ((155 - 75) X (.8) + 75 = 139) THRR: 123 - 139. Patients will then adjust their exercise intensity to match this target heart rate range for the duration of their time in cardiac rehabilitation. Cardiac rehabilitation staff will provide feedback about heart rate when they are able.
  Interventions: Behavioral: Graded Exercise Stress test (GXT) with Target Heart Rate Range
- Exercise Test, Heart Rate Range, and Heart Rate Monitor (Experimental): Patients randomly assigned to this group will also undergo a stress test (GXT) and exercise within a target heart rate range (THRR) during cardiac rehabilitation comparable to second arm of the trial. Additionally, they will receive a personal heart rate monitor (HRM). This monitor will consist of a polar heart rate chest strap and polar watch. Patients will be asked to wear this during cardiac rehabilitation and adjust their own exercise intensity. This will provide continuous feedback to the patient about their heart rate. Cardiac rehabilitation staff will also provide feedback when available.
  The investigators are using the heart rate monitors because cardiac rehab staff are not always able to adjust exercise intensity for all patients, and telemetry is not always used.
  Interventions: Behavioral: Graded Exercise Stress test (GXT) with Target Heart Rate Range; Behavioral: Heart rate monitors

INTERVENTIONS:
Behavioral: Graded Exercise Stress test (GXT) with Target Heart Rate Range — Patients assigned to one of two intervention groups will complete a GXT prior to the 4th CR session. The GXT will be completed in Baystate Medical Center's stress lab using standard protocols. This test will be used to set the target heart rate range, which will guide exercise intensity for the remainder of exercise training in cardiac rehabilitation.
  Arms: Exercise Test and Heart Rate Range; Exercise Test, Heart Rate Range, and Heart Rate Monitor
Behavioral: Heart rate monitors — Heart rate monitors (HRM) will be given to half of the patients randomly assigned to exercise stress testing group. Patients will receive a polar heart rate chest strap and polar watch. Patients will be asked to wear both, the chest strap and the watch during cardiac rehabilitation. Ultimately, we hope that the use of HRM is not necessary, but it may be needed to assure that patients in the THHR are able to consistently know their HR and adjust their exercise prescription. This will also increase the likelihood that there is a difference in heart rates between the THRR group from the RPE group.
  Arms: Exercise Test, Heart Rate Range, and Heart Rate Monitor

SUMMARY:
Cardiac Rehabilitation (CR) is an effective exercise-based lifestyle therapy for patients with cardiac disease. There are two common methods of exercise prescription, an effort based exercise prescription and target heart rate based exercise prescription. The purpose of this research study is to identify the best way to exercise in cardiac rehabilitation. There are three main goals of this study. First, the investigators want to know if an exercise test should be done near the beginning of cardiac rehabilitation. Second, the investigators want to understand what type of exercises should be recommend to patients. Third, the investigators want to understand if a personal heart rate monitor will improve adherence to a target heart rate for exercise. As part of this study, some patients will undergo an exercise stress test on a treadmill to determine a target heart rate. These patients will be given a heart rate goal to use when they exercise. Some patients will be given a personal heart rate monitor to improve adherence.

DETAILED DESCRIPTION:
Cardiac Rehabilitation (CR) is an effective exercise-based lifestyle therapy for patients with cardiac disease that reduces cardiovascular morbidity and mortality, increases quality of life, and is cost-effective. Recent retrospective studies show that higher exercise gains during CR are associated with reduced long-term morbidity and mortality among patients with both coronary artery disease and systolic heart failure. However, it is unclear which methods maximize exercise gains in CR. Recent retrospective studies have suggested that performing stress testing early in CR may allow for better tailoring of an exercise prescription and thus increase exercise gains. In this study, the investigators propose to do a randomized controlled trial of 60 patients at Baystate Medical Center CR, in which two thirds of the patients will undergo exercise testing prior to starting CR. The exercise test will determine the initial target heart rate range (THRR) and will also influence subsequent exercise progression. Additionally, half of the patients undergoing a stress test will receive a personal heart rate monitor to help improve adherence to the exercise prescription and THRR. The primary outcome is to determine feasibility, protocol fidelity, and effect sizes in preparation for a fully powered subsequent trial that will measure the impact of stress testing and a target heart rage range exercise prescription on exercise gain during CR.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are referred with an eligible diagnosis to CR.
* Patients with myocardial infarction, percutaneous coronary intervention, or bypass surgery

Exclusion Criteria:

* Permanent Atrial fibrillation, as this would interfere with using a target heart rate range during cardiac rehabilitation.
* Patients with pacemakers, as the polar heart rate monitor interferes with pacing lines on the telemetry system.
* Stable angina, as chest pain could become a limiting factor as exercise training progresses, rather than using target heart rates.
* Patients with high risk unrevascularized coronary artery disease including left main coronary disease >60% or proximal left anterior descending artery (LAD) >80%, per the discretion of the medical director.
* Patients with heart transplant or left-ventricular assist device, as heart rates can be inaccurate and difficult to measure.
* Patients who plan to attend fewer than 12 sessions of CR, for reasons that might include need to return to work, high copays, transportation, lack of insurance, or lack of interest in the program.
* Patients who join the Baystate CR program after having completed more than 3 sessions of CR at a different CR program.
* Major orthopedic limitations to exercise, such as history of amputation or exercise-limiting joint pain, or inability to walk on a treadmill, because all patients will have to complete a stress test on a treadmill and objective data collected during CR will be recorded during treadmill exercise.
* Patients who plan to undergo a clinically indicated stress test in the next 3 months as this would potentially interfere with the exercise prescription in the control group.
* Any elective hospitalization or revascularization procedure (such as PCI or CABG) that are planned to occur in the next 3 months. These could interrupt exercise training or change target heart rate ranges.
* Any other condition in which exercise training or exercise testing would be contraindicated such as severe uncontrolled hypertension, diabetes, arrhythmia, or severe valvular disease, as determined by the Medical Director of Cardiac Rehabilitation.
* Any other condition that would prohibit adherence to study protocols, such as active drug use, or untreated mental health conditions that would interfere with following instructions.
* Patients judged to be at very high or high-risk of early drop-out, per current program risk stratification

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-09-03 (Actual)

PRIMARY OUTCOMES:
Recruit 60 patients | One year
  The number of patients that signed informed consent to participate in the study
Retain patients for at least 12 exercise sessions of cardiac rehab | within 3 months of recruitment
  The percentage of patients that exercised for at least 12 sessions of cardiac rehab

SECONDARY OUTCOMES:
Peak exercise capacity at the completion of cardiac rehabilitation | Within 6 months of study enrollment
  Peak VO2 as measured on a maximal cardiopulmonary stress test
Change in functional exercise capacity from baseline to end of cardiac rehab | Within 6 months of study enrollment
  The change in functional exercise capacity as measured in METS as calculated using the online formula, http://www.fedel.com/mets/, obtained from calibrated treadmill speed and incline during usual exercise training workloads.
Adherence to Cardiac Rehabilitation (CR) | Within 6 months of enrollment
  Total number of CR sessions completed
Change in Patient Exercise Confidence | Within 6 months of enrollment
  Patients confidence, fear, and anxiety will be measured using surveys at baseline, after 6 sessions of cardiac rehab, and at the end of cardiac rehab. The confidence ruler is a 0 to 10 scale. A higher score on the confidence survey, indicates a greater level of confidence. A minimum score of 0 and a max score of 10 will be used per question, therefore, patients can receive a minimum score of 0 (low confidence) and a maximum score of 100 (high confidence). Fear and Anxiety will be measured using an anxiety questionnaire. Each question has a scale from 1 to 5 indicting very little fear to very fearful. A lower score on the anxiety scale indicates less anxiety or fear. Patients can receive a score from 6 (very little fear) to 30 (very fearful).
The number of patients with at least one or more adverse events in CR | Within 6 months of enrollment
  The percentage of patients that have an adverse clinical event that precludes or stops exercise during cardiac rehabilitation. The adverse event is determined by the opinion of the treating clinician, the patient was unable to start or continue exercising based on one or more of the following subcategories; high or low blood pressure, dyspnea, tachycardia, or chest pain as defined by the treating clinician who stopped or precluded exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Peter K Lindenauer, MD, Study Director — Baystate Medical Center
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available within 12 months of study completion.
Access Criteria: Data access requests will be reviewed by an external independent review panel. Requestors will be required to sign a data access agreement

REFERENCES:
- [Background] Heran BS, Chen JM, Ebrahim S, Moxham T, Oldridge N, Rees K, Thompson DR, Taylor RS. Exercise-based cardiac rehabilitation for coronary heart disease. Cochrane Database Syst Rev. 2011 Jul 6;(7):CD001800. doi: 10.1002/14651858.CD001800.pub2. PMID 21735386
- [Background] Brawner CA, Abdul-Nour K, Lewis B, Schairer JR, Modi SS, Kerrigan DJ, Ehrman JK, Keteyian SJ. Relationship Between Exercise Workload During Cardiac Rehabilitation and Outcomes in Patients With Coronary Heart Disease. Am J Cardiol. 2016 Apr 15;117(8):1236-41. doi: 10.1016/j.amjcard.2016.01.018. Epub 2016 Jan 28. PMID 26897640
- [Background] Keteyian SJ, Leifer ES, Houston-Miller N, Kraus WE, Brawner CA, O'Connor CM, Whellan DJ, Cooper LS, Fleg JL, Kitzman DW, Cohen-Solal A, Blumenthal JA, Rendall DS, Pina IL; HF-ACTION Investigators. Relation between volume of exercise and clinical outcomes in patients with heart failure. J Am Coll Cardiol. 2012 Nov 6;60(19):1899-905. doi: 10.1016/j.jacc.2012.08.958. Epub 2012 Oct 10. PMID 23062530
- [Background] Brawner CA, Al-Mallah MH, Ehrman JK, Qureshi WT, Blaha MJ, Keteyian SJ. Change in Maximal Exercise Capacity Is Associated With Survival in Men and Women. Mayo Clin Proc. 2017 Mar;92(3):383-390. doi: 10.1016/j.mayocp.2016.12.016. Epub 2017 Feb 6. PMID 28185659
- [Background] Keteyian SJ, Kerrigan DJ, Ehrman JK, Brawner CA. Exercise Training Workloads Upon Exit From Cardiac Rehabilitation in Men and Women: THE HENRY FORD HOSPITAL EXPERIENCE. J Cardiopulm Rehabil Prev. 2017 Jul;37(4):257-261. doi: 10.1097/HCR.0000000000000210. PMID 27755258
- [Background] Ades PA. Cardiac rehabilitation and secondary prevention of coronary heart disease. N Engl J Med. 2001 Sep 20;345(12):892-902. doi: 10.1056/NEJMra001529. No abstract available. PMID 11565523
- [Background] Suaya JA, Shepard DS, Normand SL, Ades PA, Prottas J, Stason WB. Use of cardiac rehabilitation by Medicare beneficiaries after myocardial infarction or coronary bypass surgery. Circulation. 2007 Oct 9;116(15):1653-62. doi: 10.1161/CIRCULATIONAHA.107.701466. Epub 2007 Sep 24. PMID 17893274
- [Background] Pack QR, Squires RW, Lopez-Jimenez F, Lichtman SW, Rodriguez-Escudero JP, Zysek VN, Thomas RJ. The current and potential capacity for cardiac rehabilitation utilization in the United States. J Cardiopulm Rehabil Prev. 2014 Sep-Oct;34(5):318-26. doi: 10.1097/HCR.0000000000000076. PMID 25098437
- [Background] Anderson L, Oldridge N, Thompson DR, Zwisler AD, Rees K, Martin N, Taylor RS. Exercise-Based Cardiac Rehabilitation for Coronary Heart Disease: Cochrane Systematic Review and Meta-Analysis. J Am Coll Cardiol. 2016 Jan 5;67(1):1-12. doi: 10.1016/j.jacc.2015.10.044. PMID 26764059
- [Background] Myers J, Prakash M, Froelicher V, Do D, Partington S, Atwood JE. Exercise capacity and mortality among men referred for exercise testing. N Engl J Med. 2002 Mar 14;346(11):793-801. doi: 10.1056/NEJMoa011858. PMID 11893790
- [Background] Keteyian SJ, Brawner CA, Savage PD, Ehrman JK, Schairer J, Divine G, Aldred H, Ophaug K, Ades PA. Peak aerobic capacity predicts prognosis in patients with coronary heart disease. Am Heart J. 2008 Aug;156(2):292-300. doi: 10.1016/j.ahj.2008.03.017. Epub 2008 May 22. PMID 18657659
- [Background] Pack QR, Bauldoff G, Lichtman SW, Buckley M, Eichenauer K, Gavic A, Garvey C, King ML; American Association of Cardiovascular and Pulmonary Rehabilitation Quality of Care Committee. Prioritization, Development, and Validation of American Association of Cardiovascular and Pulmonary Rehabilitation Performance Measures. J Cardiopulm Rehabil Prev. 2018 Jul;38(4):208-214. doi: 10.1097/HCR.0000000000000358. PMID 29944573
- [Background] Soga Y, Yokoi H, Ando K, Shirai S, Sakai K, Kondo K, Goya M, Iwabuchi M, Nobuyoshi M. Safety of early exercise training after elective coronary stenting in patients with stable coronary artery disease. Eur J Cardiovasc Prev Rehabil. 2010 Apr;17(2):230-4. doi: 10.1097/HJR.0b013e3283359c4e. PMID 20051870
- [Background] Iliou MC, Pavy B, Martinez J, Corone S, Meurin P, Tuppin P; CRS investigators and GERS (Groupe Exercice Readaptation, Sport) from French Society of Cardiology. Exercise training is safe after coronary stenting: a prospective multicentre study. Eur J Prev Cardiol. 2015 Jan;22(1):27-34. doi: 10.1177/2047487313505819. Epub 2013 Sep 20. PMID 24057686
- [Background] Pavy B, Iliou MC, Meurin P, Tabet JY, Corone S; Functional Evaluation and Cardiac Rehabilitation Working Group of the French Society of Cardiology. Safety of exercise training for cardiac patients: results of the French registry of complications during cardiac rehabilitation. Arch Intern Med. 2006 Nov 27;166(21):2329-34. doi: 10.1001/archinte.166.21.2329. PMID 17130385
- [Background] Hamm LF. Point: High quality or just average - the need for exercise testing before cardiac rehabilitation. Journal of Clinical Exercise Physiology. 2013;2:42-45
- [Background] McConnell TR. Counterpoint: All patients do no need an exercise test before starting cardiac rehabilitation. Journal of Clinical Exercise Physiology. 2013;2:45-48
- [Background] Scheinowitz M, Harpaz D. Safety of cardiac rehabilitation in a medically supervised, community-based program. Cardiology. 2005;103(3):113-7. doi: 10.1159/000083433. Epub 2005 Jan 19. PMID 15665529
- [Background] Goto Y, Sumida H, Ueshima K, Adachi H, Nohara R, Itoh H. Safety and implementation of exercise testing and training after coronary stenting in patients with acute myocardial infarction. Circ J. 2002 Oct;66(10):930-6. doi: 10.1253/circj.66.930. PMID 12381088
- [Background] Fletcher GF, Balady GJ, Amsterdam EA, Chaitman B, Eckel R, Fleg J, Froelicher VF, Leon AS, Pina IL, Rodney R, Simons-Morton DA, Williams MA, Bazzarre T. Exercise standards for testing and training: a statement for healthcare professionals from the American Heart Association. Circulation. 2001 Oct 2;104(14):1694-740. doi: 10.1161/hc3901.095960. No abstract available. PMID 11581152
- [Derived] Shea MG, Headley S, Mullin EM, Brawner CA, Schilling P, Pack QR. Comparison of Ratings of Perceived Exertion and Target Heart Rate-Based Exercise Prescription in Cardiac Rehabilitation: A RANDOMIZED CONTROLLED PILOT STUDY. J Cardiopulm Rehabil Prev. 2022 Sep 1;42(5):352-358. doi: 10.1097/HCR.0000000000000682. Epub 2022 Mar 31. PMID 35383680